CLINICAL TRIAL: NCT02148523
Title: Using Social Comparison To Improve Medication Adherence In Statin Users With Diabetes
Brief Title: Social Forces to Improve Statin Adherence (Study B)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 819129-B
Record Dates: First submitted 2013-12-17; First posted 2014-05-28 (Estimated); Results first posted 2017-05-23 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Medication Adherence; High Blood Pressure; Diabetes
Keywords: Medication Adherence; High Blood Pressure; Diabetes; Statins
MeSH Terms: conditions — Medication Adherence; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Weekly Adherence Report (Experimental): Adherence report to subject every 7 days.
  Interventions: Behavioral: Adherence feedback; Device: Electronic pill bottle
- Weekly Adherence Peer-Comparison Report (Experimental): Adherence report to subject every 7 days with tailored comparison messages based on subject's adherence.
  Interventions: Behavioral: Comparison to peers; Device: Electronic pill bottle
- Usual Care (Other): Usual care with GlowCap.
  Interventions: Device: Electronic pill bottle

INTERVENTIONS:
Behavioral: Comparison to peers
  Arms: Weekly Adherence Peer-Comparison Report
Behavioral: Adherence feedback
  Arms: Weekly Adherence Report
Device: Electronic pill bottle — This device can remotely track medication taking and will be used by subjects to store once-a-day statin medication already prescribed pre-trial.
  Other Names: Vitality GlowCap

SUMMARY:
To assess the effectiveness of social comparison in improving the outcome of statin adherence versus usual care as measured by an electronic pill bottle.

Subjects receiving weekly reports with their adherence and information about their place in the distribution of their peers will have the highest statin adherence of any arm, as measured by electronic pill bottle.

DETAILED DESCRIPTION:
We propose to complete a randomized controlled trial (RCT) of 201 subjects with medication treated diabetes and evidence of poor adherence to a statin medication (<70% medication possession ratio (MPR) determined through pharmacy records; no combination meds). Study subjects will use GlowCaps to store their statin medication.

Arm 1 will receive weekly feedback containing general information about the subject's adherence (i.e., reminding the subject how many days that week he or she took the medication). Arm 2 will be provided the same weekly feedback and the information of whether his or her adherence is above or below the average adherence in their arm, along with a message of encouragement tailored to their place in the arm distribution. Subjects with perfect adherence will receive: "You took your pill every day for the last 7 days. Great job! Keep it up" with their weekly adherence report. Subjects with less than perfect adherence and adherence rate in the top 50% of the arm will receive: "You took your pill for ** days out of the last 7 days. Your medication adherence was as good or better than half of people in this study. Taking your pill every day would improve your health even more" with their weekly adherence report. Subjects with less than perfect adherence and adherence rate in the bottom 50% of the arm will receive: "You took your pill for ** days out of the last 7 days. Your medication adherence was in the bottom half of the people in this study. If you took your pill more often, you could be in the top half of people in the study" with their weekly adherence report. Adherence records will be displayed on each subject's Way to Health (WTH) account in all arms. Arm 3 will be the usual care control.

ELIGIBILITY:
Inclusion Criteria:

* The subject is Humana insured
* The subject is an English speaking adult
* Age range ≥18 years
* The subject has diagnosis with diabetes for ≥12 months
* The subject has an MPR <70% to a statin medication
* Subjects denies side-effects to their statin medication

Exclusion Criteria:

* The subject is <18 years old
* The subject is considered part of a vulnerable population (is a prisoner, a cognitively impaired person, or a pregnant woman)
* On statin combination medication
* The subject does not identify an individual who agrees to serve as their MAP
* The subject reports a clinically important side effect to the statin medication or active liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter P Reese, MD, MSCE, Principal Investigator — UPenn, PSOM; Judd B Kessler, PhD, Principal Investigator — UPenn, Wharton; Kevin Volpp, MD, PhD, Principal Investigator — UPenn, PSOM
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Weekly Adherence Report: Adherence report to subject every 7 days.
  Adherence feedback
  Electronic pill bottle: This device can remotely track medication taking and will be used by subjects to store once-a-day statin medication already prescribed pre-trial.
- Weekly Adherence Peer-Comparison Report: Adherence report to subject every 7 days with tailored comparison messages based on subject's adherence.
  Comparison to peers
  Electronic pill bottle: This device can remotely track medication taking and will be used by subjects to store once-a-day statin medication already prescribed pre-trial.
Period: Overall Study
Arm/Group | Weekly Adherence Report | Weekly Adherence Peer-Comparison Report | Usual Care
Started | 67 | 67 | 67
Completed | 67 | 67 | 67
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Weekly Adherence Report | Weekly Adherence Peer-Comparison Report | Usual Care | Total
Number analyzed (Participants) | 67 | 67 | 67 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (11) | 68 (10) | 67 (10) | 67 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 25 | 28 | 87
  Male | 33 | 42 | 39 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 2 | 8
  Not Hispanic or Latino | 65 | 63 | 65 | 193
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 3 | 1 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 8 | 2 | 18
  White | 54 | 56 | 63 | 173
  More than one race | 2 | 1 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Statin Adherence
Description: The primary outcome will be the percent of statin doses taken during the study as measured by the GlowCaps.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: percentage of correct statin doses
Arm/Group | Weekly Adherence Report | Weekly Adherence Peer-Comparison Report | Usual Care
Number analyzed (Participants) | 67 | 67 | 67
percentage of correct statin doses | 79 (.26) | 84 (.23) | 80 (.23)

2. Secondary Outcome: Morisky Medication Adherence Scale (MMAS)
Description: The secondary outcome will be subjects' self-reports medication adherence. Morisky et al. developed this 8-item MMAS (MMAS-8) in 2008. The first seven items are Yes/No responses while the last item is a 5-point Likert response. The scoring scheme is: "Yes" = 0 and "No" = 1 (and "0" = 0 and "1-4" = 1 for Likert question). The items are summed to give a range of scores from 0 to 8. Respondents' summed score get grouped as follows: "0" = High Adherence; "1-2" = Medium Adherence; "3-8" = Low Adherence.
Time Frame: 90 days
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Weekly Adherence Report | Weekly Adherence Peer-Comparison Report | Usual Care
Number analyzed (Participants) | 67 | 67 | 67
units on a scale | 6 [4.75 to 7] | 6 [5 to 7] | 5.5 [4.75 to 7]

ADVERSE EVENTS:
Arm/Group | Weekly Adherence Report | Weekly Adherence Peer-Comparison Report | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/67 | 0/67
Other Adverse Events (participants affected / at risk) | 0/67 | 0/67 | 0/67

LIMITATIONS AND CAVEATS:
The interventions lasted only 3 months; differences in adherence might emerge over a longer period of time. The primary outcome of pill-bottle-measured adherence has limitations, including bottle malfunction.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No